CLINICAL TRIAL: NCT06279871
Title: A Phase 3, Multicenter, Observer-blind, Randomized, Controlled Study to Evaluate the Immunogenicity, Reactogenicity, and Safety of a Self-Amplifying RNA COVID-19 Vaccine (ARCT-2303), Administered Concomitantly With Quadrivalent Influenza Vaccines, in Adults
Brief Title: Immunogenicity and Safety Study of Self-amplifying mRNA COVID-19 Vaccine Administered With Influenza Vaccines in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Collaborators: Seqirus (Industry); Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARCT-2303-01
Record Dates: First submitted 2024-02-23; First posted 2024-02-28 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1a (ARCT-2303/Influenza vaccine) (Experimental): Participants will receive one 0.5-mL IM (intramuscular) dose of ARCT-2303 and one 0.5-mL IM dose of influenza vaccine on Day 1 followed by a 0.5-mL IM dose of placebo on Day 29.
  Interventions: Biological: ARCT-2303; Biological: Influenza vaccine; Other: Placebo
- Group 2a (ARCT-2303) (Experimental): Participants will receive one 0.5-mL IM dose of ARCT-2303 and one 0.5-mL IM dose of placebo on Day 1 followed by a 0.5-mL IM dose of influenza vaccine on Day 29.
  Interventions: Biological: ARCT-2303; Biological: Influenza vaccine; Other: Placebo
- Group 3a (Influenza vaccine) (Active Comparator): Participants will receive one 0.5-mL IM dose of influenza vaccine and one 0.5-mL IM dose of placebo on Day 1 followed by a 0.5-mL IM dose of ARCT-2303 on Day 29.
  Interventions: Biological: ARCT-2303; Biological: Influenza vaccine; Other: Placebo
- Group 1b (ARCT-2303/ Influenza vaccine) (Experimental): Participants will receive one 0.5-mL IM dose of ARCT-2303 and one 0.5-mL IM dose of influenza vaccine on Day 1 followed by a 0.5-mL IM dose of placebo on Day 29.
  Interventions: Biological: ARCT-2303; Biological: Influenza vaccine, adjuvanted; Other: Placebo
- Group 2b (ARCT-2303) (Experimental): Participants will receive one 0.5-mL IM dose of ARCT-2303 and one 0.5-mL IM dose of placebo on Day 1 followed by a 0.5-mL IM dose of influenza vaccine on Day 29.
  Interventions: Biological: ARCT-2303; Biological: Influenza vaccine, adjuvanted; Other: Placebo
- Group 3b (Influenza vaccine) (Active Comparator): Participants will receive one 0.5-mL IM dose of influenza vaccine and one 0.5-mL IM dose of placebo on Day 1 followed by a 0.5-mL IM dose of ARCT-2303 on Day 29.
  Interventions: Biological: ARCT-2303; Biological: Influenza vaccine, adjuvanted; Other: Placebo

INTERVENTIONS:
Biological: ARCT-2303 — Self-Amplifying RNA COVID-19 vaccine (Omicron XBB.1.5)
Biological: Influenza vaccine — Licensed cell-based influenza vaccine
  Arms: Group 1a (ARCT-2303/Influenza vaccine); Group 2a (ARCT-2303); Group 3a (Influenza vaccine)
Biological: Influenza vaccine, adjuvanted — Licensed influenza vaccine, adjuvanted
  Arms: Group 1b (ARCT-2303/ Influenza vaccine); Group 2b (ARCT-2303); Group 3b (Influenza vaccine)
Other: Placebo — 0.9% saline

SUMMARY:
This is a multicenter, observer-blind, randomized, controlled phase 3 study to evaluate the immunogenicity, reactogenicity, and safety of an investigational self-amplifying RNA COVID-19 vaccine (ARCT-2303) administered concomitantly with quadrivalent influenza vaccines or standalone in adults who previously received authorized COVID-19 vaccine.

DETAILED DESCRIPTION:
Approximately 1680 participants previously vaccinated with authorized COVID-19 vaccine will be enrolled in this study in two age cohorts (younger adults and older adults). Within each cohort, participants will be randomly assigned in a ratio of 1:1:1 to receive the ARCT-2303 vaccine concomitantly with a quadrivalent influenza vaccine, the ARCT-2303 vaccine and placebo, or the quadrivalent influenza vaccine and placebo. The assessment of immunogenicity will be performed 28 days after vaccination. To provide equal benefit from the participation in the study and complete seasonal vaccination against COVID-19 and influenza, a switchover vaccine dose (influenza, ARCT-2303 or placebo) will be administered 28 days after initial vaccination. All participants will be followed up for safety assessment until the end of the study.

A historical control group vaccinated on a similar schedule (ARCT-154 vaccine) from a previous study (ARCT-154-J01) will be used to compare with the immunogenicity of the ARCT-2303 vaccine.

Cohort A (younger adults; approximately 1200 participants):

* Group 1a (ARCT-2303/Influenza vaccine): participants will receive one dose of ARCT-2303 and one dose of Influenza vaccine (opposite arms) on Day 1, and one dose of placebo on Day 29.
* Group 2a (ARCT-2303): participants will receive one dose of ARCT-2303 and one dose of placebo (opposite arms) on Day 1, and one dose of Influenza vaccine on Day 29.
* Group 3a (Influenza vaccine): participants will receive one dose of Influenza vaccine and one dose of placebo (opposite arms) on Day 1, and one dose of ARCT-2303 on Day 29.

Cohort B (older adults; approximately 480 participants):

* Group 1b (ARCT-2303/Influenza vaccine): participants will receive one dose of ARCT-2303 and one dose of Influenza vaccine (opposite arms) on Day 1, and one dose of placebo on Day 29.
* Group 2b (ARCT-2303): participants will receive one dose of ARCT-2303 and one dose of placebo (opposite arms) on Day 1, and one dose of Influenza vaccine on Day 29.
* Group 3b (Influenza vaccine): participants will receive one dose of Influenza vaccine and one dose of placebo (opposite arms) on Day 1, and one dose of ARCT-2303 on Day 29.

ELIGIBILITY:
Inclusion Criteria:

1, Individuals are male, female, or transgender adults ≥18 years of age.

2. Healthy participants or participants with pre-existing stable medical conditions.

3. Participant or legally authorized representatives must freely provide documented informed consent prior to study procedures being performed.

4. Individuals must have been previously vaccinated with COVID-19 vaccines.

5. Individuals of childbearing potential must be willing to adhere to contraceptive requirements.

Exclusion Criteria:

1. Individuals with acute medical illness or febrile illness.
2. Individuals with a positive SARS-CoV-2 rapid antigen test at Screening.
3. Individuals with a history of COVID-19 or virologically confirmed SARS-CoV-2 infection within the past 5 months or history of COVID-19 with ongoing sequelae.
4. Individuals with a known history of severe hypersensitivity reactions, including anaphylaxis, or other significant adverse reactions to any components of mRNA vaccine, or influenza vaccine, including egg protein.
5. Individuals who have a positive pregnancy test at the Screening visit or who intend to become pregnant or breastfeed during the study.
6. Individuals with a history of myocarditis, pericarditis, myopericarditis or cardiomyopathy.
7. Individuals with a history of Guillain-Barré syndrome, encephalomyelitis, or transverse myelitis.
8. Individuals with a history of congenital or acquired immunodeficiency.
9. Individuals who have received immunomodulatory, immunostimulatory, or immunosuppressant drugs within 3 months of Screening; or individuals requiring systemic corticosteroids exceeding 10 mg/day of prednisone equivalent for ≥10 days within 30 days of Screening.
10. Individuals who have received immunoglobulins and/or any blood or blood products within the 3 months before the first vaccine administration or plan to receive such products at any time during the study.
11. Individuals with a documented history of HIV infection, or who are currently known to have active tuberculosis.
12. Individuals receiving treatment with another investigational drug, biological agent, or device.
13. Individuals who have received any investigational COVID-19 vaccines.
14. Individuals who received any influenza vaccine within 6 months prior to enrollment or plan to receive an influenza vaccine during the study period.
15. Individuals who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to 14 days after the study vaccination.
16. Individuals who are investigator site staff members, employees of the Sponsor or the Clinical Research Organization directly involved in the conduct of the study, or site staff members otherwise supervised by the investigator or immediate family members of any of the previously mentioned individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1514 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Arcturus Therapeutics
Locations (29):
- Australia (22):
  - Paratus Clinical Canberra, Canberra, Australian Capital Territory
  - Paratus Clinical Central Coast, Central Coast, New South Wales
  - Sutherland Shire Clinical Research - Walski, Miranda, New South Wales
  - Australian Clinical Research Network (ACRN), Sydney, New South Wales
  - Austrials - St. Leonards, Sydney, New South Wales
  - Emeritus Research Sydney, Sydney, New South Wales
  - Griffith University Clinical Trials Unit, Sydney, New South Wales
  - Northern Beaches Clinical Research - Walski, Sydney, New South Wales
  - Paratus Clinical Blacktown, Sydney, New South Wales
  - Wollongong Clinical Research, Wollongong, New South Wales
  - Nucleus Network Brisbane (Q-Pharm), Brisbane, Queensland
  - Paratus Clinical Brisbane, Brisbane, Queensland
  - USC Southbank, Brisbane, Queensland
  - USC Morayfield, Morayfield, Queensland
  - USC Sippy Down, Sunshine Coast, Queensland
  - CMAX, Adelaide, South Australia
  - Austrials -Sunshine, Melbourne, Victoria
  - Emeritus Research Melbourne, Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria
  - The Peter Doherty Institute for Infection and Immunity, Melbourne, Victoria
  - Veritus Research, Melbourne, Victoria
  - Clinitrials - Mount Site, Perth, Western Australia
- Costa Rica (2):
  - Clínica San Agustín, San José
  - IICIMED, San José
- Honduras (3):
  - Organización y centro de investigación clínica Ochoa (OCINCO), Comayagua
  - Deposito de Medicamentos de Investigación Cousin Agustín (DEMEDICA), San Pedro Sula
  - Inversiones en Investigación Médica S.A (INVERIME), Tegucigalpa
- Philippines (2):
  - Tropical Disease Foundation - Putatan Health Center, City of Muntinlupa
  - Far Eastern University - Nicanor R. M Foundation, Quezon City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giles ML, Tabora C, Baccarini C, Barrientos L, Vargas JC, Montellano ME, Nguyen P, Deshmukh S, Neville M, Hohenboken M, van Boxmeer J, Jin H, Bugarini R, Liu X, Walson JL, Verhoeven C, Smolenov I. Immunogenicity and safety of self-amplifying mRNA COVID-19 vaccine (ARCT-2303), with or without co-administration of seasonal inactivated influenza vaccine in adults: a phase 3, randomised, controlled, observer-blind, multicentre study. EClinicalMedicine. 2025 Aug 20;87:103428. doi: 10.1016/j.eclinm.2025.103428. eCollection 2025 Sep. PMID 40896462

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study utilized the study group (ARCT-154 vaccine) from study ARCT-154-J01 as a historical control. The participants in the historical control arm were not considered enrolled in this study.
Groups:
- Cohort A Group 1a: ARCT-2303+ Quadrivalent Influenza Vaccine (QIV) + Placebo: Younger adult participants received one dose of ARCT-2303 and one dose of QIV on Day 1, and one dose of placebo on Day 29.
- Cohort A Group 2a: ARCT-2303 + Placebo + QIV: Younger adult participants received one dose of ARCT-2303 and one dose of placebo on Day 1, and one dose of QIV on Day 29.
- Cohort A Group 3a: QIV + Placebo + ARCT-2303: Younger adult participants received one dose of QIV and one dose of placebo on Day 1, and one dose of ARCT-2303 on Day 29.
- Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo: Older adult participants received one dose of ARCT-2303 and one dose of aQIV on Day 1, and one dose of placebo on Day 29.
- Cohort B Group 2b: ARCT-2303 + Placebo + aQIV: Older adult participants received one dose of ARCT-2303 and one dose of placebo on Day 1, and one dose of aQIV on Day 29.
- Cohort B Group 3b: aQIV + Placebo + ARCT-2303: Older adult participants received one dose of aQIV and one dose of placebo on Day 1, and one dose of ARCT-2303 on Day 29.
- ARCT-154-J01 (Historical Control): Participants from study ARCT-154-J01 with available pre- and post-vaccination serum samples who were allocated in the ARCT-154 group. This group of participants was used as a historical control group.
Period: Overall Study
Arm/Group | Cohort A Group 1a: ARCT-2303+ Quadrivalent Influenza Vaccine (QIV) + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV | Cohort A Group 3a: QIV + Placebo + ARCT-2303 | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV | Cohort B Group 3b: aQIV + Placebo + ARCT-2303 | ARCT-154-J01 (Historical Control)
Started | 408 | 406 | 405 | 99 | 98 | 98 | 385
Received Dose 1 | 403 | 403 | 398 | 99 | 98 | 98 | 385 (Number of participants who received study drug in the historical control study.)
Received Dose 2 | 393 | 394 | 390 | 95 | 97 | 96 | 0
Completed | 392 | 387 | 389 | 97 | 98 | 97 | 385
Not Completed | 16 | 19 | 16 | 2 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other than Specified | 1 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 4 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 11 | 10 | 8 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT), all participants who received at least one dose of a study vaccine in this study. Data are also reported for participants from study ARCT-154-J01 (historical control group), which included participants from ARCT-154-J01 who received ARCT-154 booster vaccine, provided evaluable pre-/post-vaccination blood samples, and did not have SARS-CoV-2 infection/protocol deviations that impacted immunogenicity assessment. Participants were analyzed according to the vaccine assigned.
Groups:
- Cohort A Group 1a: ARCT-2303+ QIV + Placebo: Younger adult participants received one dose of ARCT-2303 and one dose of QIV on Day 1, and one dose of placebo on Day 29.
- Total: Total of all reporting groups
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV | Cohort A Group 3a: QIV + Placebo + ARCT-2303 | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV | Cohort B Group 3b: aQIV + Placebo + ARCT-2303 | ARCT-154-J01 (Historical Control) | Total
Number analyzed (Participants) | 403 | 403 | 398 | 99 | 98 | 98 | 385 | 1884
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (12.0) | 36.8 (12.1) | 39.2 (11.9) | 69.6 (5.3) | 70.4 (5.4) | 70.4 (4.9) | 45.3 (11.9) | 44.2 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 255 | 243 | 64 | 68 | 63 | 228 | 1180
  Male | 144 | 148 | 155 | 35 | 30 | 35 | 157 | 704
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65 | 67 | 64 | 23 | 15 | 21 | 0 | 255
  Not Hispanic or Latino | 333 | 333 | 332 | 76 | 83 | 77 | 385 | 1619
  Unknown or Not Reported | 5 | 3 | 2 | 0 | 0 | 0 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 11 | 16 | 4 | 6 | 5 | 0 | 60
  Asian | 150 | 159 | 177 | 69 | 77 | 68 | 385 | 1085
  Native Hawaiian or Other Pacific Islander | 7 | 3 | 2 | 0 | 0 | 0 | 0 | 12
  Black or African American | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 3
  White | 179 | 173 | 158 | 9 | 8 | 10 | 0 | 537
  More than one race | 14 | 15 | 13 | 7 | 2 | 3 | 0 | 54
  Unknown or Not Reported | 34 | 42 | 30 | 10 | 5 | 12 | 0 | 133

OUTCOME MEASURES:

1. Primary Outcome: Groups 2a and 2b and ARCT-154-J01 Historical Control: Geometric Mean Titers (GMT) of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Neutralizing Antibody Titers Against Omicron XBB.1.5 Subvariant at Day 29
Time Frame: Day 29
Population: Study treatment arm: per protocol (PP) set for immunogenicity, participants in the Modified Intent-To-Treat Analysis Set (mITT) who correctly received all protocol-required doses of study vaccines at Day 1 and who at or prior to the specified timepoint (Day 29 or Day 181) had no evidence of SARS-CoV-2 infection and no protocol deviations impacting the analysis of immunogenicity data. As pre-specified, data for groups 2a & 2b were collected and are reported pooled as a combined group.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Cohort A Group 2a: ARCT-2303 + Placebo + QIV and Cohort B Group 2b: ARCT-2303 + Placebo + aQIV: Cohort A Group 2a: Younger adult participants received one dose of ARCT-2303 and one dose of placebo on Day 1, and one dose of QIV on Day 29. Cohort B Group 2b: Older adult participants received one dose of ARCT-2303 and one dose of placebo on Day 1, and one dose of aQIV on Day 29.
Arm/Group | Cohort A Group 2a: ARCT-2303 + Placebo + QIV and Cohort B Group 2b: ARCT-2303 + Placebo + aQIV | ARCT-154-J01 (Historical Control)
Number analyzed (Participants) | 473 | 385
Titer | 718 [652 to 791] | 263 [236 to 293]

2. Primary Outcome: Groups 2a and 2b and ARCT-154-J01 Historical Control: Number of Participants With Seroconversion to SARS-CoV-2 Neutralizing Antibody Against Omicron XBB.1.5 Subvariant at Day 29
Description: Seroconversion was defined as either a pre-vaccination titer below the lower limit of quantitation (LLOQ) and a postvaccination titer ≥4xLLOQ; or a pre-vaccination titer ≥LLOQ and a ≥4-fold increase in post-vaccination titer.
Time Frame: Day 29
Population: Study treatment arm: PP set for immunogenicity, which included participants in the mITT who correctly received all protocol-required doses of study vaccines at Day 1 and who at or prior to the specified timepoint (Day 29) had no evidence of SARS-CoV-2 infection and no protocol deviations impacting the analysis of immunogenicity data. As pre-specified, data for groups 2a &2b were collected and are reported pooled as a combined group.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Group 2a: ARCT-2303 + Placebo + QIV and Cohort B Group 2b: ARCT-2303 + Placebo + aQIV | ARCT-154-J01 (Historical Control)
Number analyzed (Participants) | 473 | 385
Participants | 349 | 175

3. Primary Outcome: Groups 1a and 3a: Adjusted Hemagglutination Inhibition (HI) GMTs Against Influenza Vaccine Strains at Day 29
Description: Influenza vaccine strains were A/H1N1, A/H3N2, B/Victoria, and B/Yamagata.
Time Frame: Day 29
Population: PP set for immunogenicity, which included participants in the mITT who correctly received all protocol-required doses of study vaccines at Day 1 and who at or prior to the specified timepoint (Day 29) had no evidence of SARS-CoV-2 infection and no protocol deviations impacting the analysis of immunogenicity data.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 3a: QIV + Placebo + ARCT-2303
Number analyzed (Participants) | 375 | 376
titers
  A/H1N1 | 338 [289 to 395] | 354 [304 to 413]
  A/H3N2 | 280 [242 to 325] | 269 [232 to 311]
  B/Victoria | 109 [92 to 129] | 99 [84 to 117]
  B/Yamagata | 123 [111 to 137] | 112 [101 to 125]

4. Primary Outcome: Groups 1a and 2a: Adjusted GMTs of SARS-CoV-2 Neutralizing Antibody Against Omicron XBB.1.5 Subvariant at Day 29
Time Frame: Day 29
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV
Number analyzed (Participants) | 375 | 378
titers | 768 [680 to 867] | 954 [844 to 1077]

5. Secondary Outcome: Groups 1a and 2a: GMT of SARS-CoV-2 Neutralizing Antibodies Against Omicron XBB.1.5 Subvariant at Days 1, 29 and 181
Time Frame: Group 1a: Days 1 and 29; Group 2a: Days 1, 29, and 181
Population: PP set for immunogenicity, which included participants in the mITT who correctly received all protocol-required doses of study vaccines at Day 1 and who at or prior to the specified timepoint (Day 29 or Day 181) had no evidence of SARS-CoV-2 infection and no protocol deviations impacting the analysis of immunogenicity data. Overall number of participants analyzed = participants evaluable for this outcome measure. Number analyzed = participants evaluable at the specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV
Number analyzed (Participants) | 375 | 378
titers
  Day 1 | 118 [103 to 135] | 140 [123 to 169]
  Day 29 | 789 [708 to 880] | 1072 [957 to 1199]
  Day 181: number analyzed (Participants) | 0 | 93
  Day 181 |  | 794 [653 to 967]

6. Secondary Outcome: Groups 1a and 2a: Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Neutralizing Antibodies Against Omicron XBB.1.5 Subvariant at Days 29 and 181
Description: GMFR is reported as a ratio to Day 1.
Time Frame: Group 1a: Day 29; Group 2a: Days 29 and 181
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV
Number analyzed (Participants) | 375 | 378
ratio
  Day 29 | 6.7 [6.0 to 7.5] | 7.7 [6.8 to 8.6]
  Day 181: number analyzed (Participants) | 0 | 93
  Day 181 |  | 5.3 [4.2 to 6.7]

7. Secondary Outcome: Groups 1a and 2a: Number of Participants With Seroconversion of SARS-CoV-2 Neutralizing Antibodies Against Omicron XBB.1.5 Subvariant at Day 29
Description: Seroconversion was defined as either a pre-vaccination titer below the LLOQ and a postvaccination titer ≥4xLLOQ; or a pre-vaccination titer ≥LLOQ and a ≥4-fold increase in post-vaccination titer.
Time Frame: Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV
Number analyzed (Participants) | 375 | 378
Participants | 242 | 279

8. Secondary Outcome: Groups 1a and 2a: Number of Participants With SARS-CoV-2 Neutralizing Antibody Against Omicron XBB.1.5 Subvariant Titer ≥ LLOQ at Days 1 and 29
Time Frame: Days 1 and 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV
Number analyzed (Participants) | 375 | 378
Participants
  Day 1 | 331 | 344
  Day 29 | 375 | 378

9. Secondary Outcome: Groups 1a and 3a: GMTs of HI Assay Titers Against Influenza Vaccine Strains at Days 1 and 29
Description: Vaccine strains were A/H1N1, A/H3N2, B/Victoria, and B/Yamagata.
Time Frame: Days 1 and 29
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 3a: QIV + Placebo + ARCT-2303
Number analyzed (Participants) | 375 | 376
titer
  A/H1N1 Day 1 | 38 [33 to 44] | 37 [32 to 43]
  A/H1N1 Day 29 | 429 [374 to 493] | 433 [381 to 491]
  A/H3N2 Day 1 | 32 [28 to 37] | 36 [31 to 42]
  A/H3N2 Day 29 | 331 [291 to 378] | 334 [295 to 377]
  B/Victoria Day 1 | 13 [12 to 15] | 15 [13 to 17]
  B/Victoria Day 29 | 109 [95 to 125] | 102 [90 to 117]
  B/Yamagata Day 1 | 29 [26 to 32] | 34 [30 to 37]
  B/Yamagata Day 29 | 132 [119 to 145] | 126 [115 to 138]

10. Secondary Outcome: Groups 1a and 3a: GMFR of HI Assay Titers Against Influenza Vaccine Strains at Day 29
Description: Vaccine strains were A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. GMFR is reported as a ratio to Day 1.
Time Frame: Day 29
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 3a: QIV + Placebo + ARCT-2303
Number analyzed (Participants) | 375 | 376
ratio
  A/H1N1 | 11.2 [9.6 to 13.2] | 11.6 [9.8 to 13.6]
  A/H3N2 | 10.3 [8.9 to 11.9] | 9.2 [8.0 to 10.6]
  B/Victoria | 8.1 [7.0 to 9.4] | 6.9 [6.0 to 7.9]
  B/Yamagata | 4.6 [4.1 to 5.1] | 3.7 [3.4 to 4.1]

11. Secondary Outcome: Groups 1a and 3a: Number of Participants With Seroconversion of HI Assay Titers Against Influenza Vaccine Strains at Day 29
Description: Seroconversion was defined as either a pre-vaccination titer below the LLOQ and a postvaccination titer ≥4xLLOQ; or a pre-vaccination titer ≥LLOQ and a ≥4-fold increase in post-vaccination titer. Vaccine strains were A/H1N1, A/H3N2, B/Victoria, and B/Yamagata.
Time Frame: Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 3a: QIV + Placebo + ARCT-2303
Number analyzed (Participants) | 375 | 376
Participants
  A/H1N1 | 267 | 259
  A/H3N2 | 266 | 266
  B/Victoria | 233 | 215
  B/Yamagata | 197 | 167

12. Secondary Outcome: Groups 1a and 3a: Number of Participants With HI Titer ≥1:40 at Days 1 and 29
Description: Vaccine strains were A/H1N1, A/H3N2, B/Victoria, and B/Yamagata.
Time Frame: Days 1 and 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 3a: QIV + Placebo + ARCT-2303
Number analyzed (Participants) | 375 | 376
Participants
  A/H1N1 Day 1 | 197 | 195
  A/H1N1 Day 29 | 354 | 367
  A/H3N2 Day 1 | 178 | 200
  A/H3N2 Day 29 | 361 | 364
  B/Victoria Day 1 | 73 | 83
  B/Victoria Day 29 | 299 | 294
  B/Yamagata Day 1 | 165 | 201
  B/Yamagata Day 29 | 345 | 347

13. Secondary Outcome: Groups 1b and 2b: GMTs of SARS-CoV-2 Neutralizing Antibodies Against Omicron XBB.1.5 Subvariant at Days 1, 29 and 181
Time Frame: Group 1b: Days 1 and 29, Group 2b: Days 1, 29 and 181
Population: PP set for immunogenicity, which included participants in the mITT who correctly received all protocol-required doses of study vaccines at Day 1 and who at or prior to the specified timepoint (Day 29 or Day 181) had no evidence of SARS-CoV-2 infection and no protocol deviations impacting the analysis of immunogenicity data. Overall number of participants analyzed = number evaluable for the outcome measure. Number analyzed = participants evaluable at the specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV
Number analyzed (Participants) | 92 | 95
titer
  Day 1 | 138 [106 to 180] | 206 [158 to 269]
  Day 29 | 932 [742 to 1170] | 1420 [1126 to 1791]
  Day 181: number analyzed (Participants) | 0 | 93
  Day 181 |  | 878 [738 to 1045]

14. Secondary Outcome: Groups 1b and 2b: GMFRs of SARS-CoV-2 Neutralizing Antibodies Against Omicron XBB.1.5 Subvariant at Days 29 and 181
Description: GMFR is reported as a ratio to Day 1.
Time Frame: Group 1b: Day 29 and Group 2b: Days 29 and 181
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV
Number analyzed (Participants) | 92 | 95
ratio
  Day 29 | 6.8 [5.3 to 8.6] | 6.9 [5.4 to 8.8]
  Day 181: number analyzed (Participants) | 0 | 93
  Day 181 |  | 4.3 [3.2 to 5.7]

15. Secondary Outcome: Groups 1b and 2b: Number of Participants With Seroconversion of SARS-CoV-2 Neutralizing Antibodies Against Omicron XBB.1.5 Subvariant at Day 29
Description: as for outcome 7
Time Frame: Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV
Number analyzed (Participants) | 92 | 95
Participants | 66 | 70

16. Secondary Outcome: Groups 1b and 2b: Number of Participants With SARS-CoV-2 Neutralizing Antibody Against Omicron XBB.1.5 Subvariant Titer ≥ LLOQ at Days 1 and 29
Time Frame: Days 1 and 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV
Number analyzed (Participants) | 92 | 95
Participants
  Day 1 | 84 | 90
  Day 29 | 92 | 95

17. Secondary Outcome: Groups 1b and 3b: GMTs of HI Assay Titers Against Influenza Vaccine Strains at Days 1 and 29
Description: Vaccine strains were A/H1N1, A/H3N2, B/Victoria, and B/Yamagata.
Time Frame: Days 1 and 29
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 3b: aQIV + Placebo + ARCT-2303
Number analyzed (Participants) | 92 | 93
titers
  A/H1N1 Day 1 | 115 [83 to 160] | 109 [78 to 153]
  A/H1N1 Day 29 | 1064 [827 to 1369] | 961 [773 to 1194]
  A/H3N2 Day 1 | 78 [56 to 110] | 92 [68 to 127]
  A/H3N2 Day 29 | 475 [368 to 613] | 453 [342 to 600]
  B/Victoria Day 1 | 20 [15 to 26] | 29 [20 to 41]
  B/Victoria Day 29 | 121 [91 to 160] | 132 [98 to 178]
  B/Yamagata Day 1 | 25 [19 to 34] | 27 [20 to 35]
  B/Yamagata Day 29 | 138 [108 to 176] | 132 [102 to 170]

18. Secondary Outcome: Groups 1b and 3b: GMFRs of of HI Assay Titers Against Influenza Vaccine Strains at Day 29
Description: Vaccine strains were A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. GMFR is reported as a ratio to Day 1.
Time Frame: Day 29
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 3b: aQIV + Placebo + ARCT-2303
Number analyzed (Participants) | 92 | 93
ratio
  A/H1N1 | 9.2 [6.4 to 13.4] | 8.8 [6.1 to 12.6]
  A/H3N2 | 6.0 [4.4 to 8.4] | 4.9 [3.6 to 6.7]
  B/Victoria | 6.2 [4.4 to 8.5] | 4.6 [3.4 to 6.1]
  B/Yamagata | 5.5 [4.0 to 7.6] | 5.0 [3.8 to 6.5]

19. Secondary Outcome: Groups 1b and 3b: Number of Participants With Seroconversion of HI Assay Titers Against Influenza Vaccine Strains at Day 29
Description: as for outcome 11
Time Frame: Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 3b: aQIV + Placebo + ARCT-2303
Number analyzed (Participants) | 92 | 93
Participants
  A/H1N1 | 59 | 59
  A/H3N2 | 50 | 42
  B/Victoria | 47 | 45
  B/Yamagata | 48 | 47

20. Secondary Outcome: Groups 1b and 3b: Number of Participants With HI Titer ≥1:40 at Days 1 and 29
Description: Vaccine strains analyzed for this outcome measure were A/H1N1, A/H3N2, B/Victoria, and B/Yamagata.
Time Frame: Days 1 and 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 3b: aQIV + Placebo + ARCT-2303
Number analyzed (Participants) | 92 | 93
Participants
  A/H1N1 Day 1 | 75 | 71
  A/H1N1 Day 29 | 92 | 93
  A/H3N2 Day 1 | 62 | 70
  A/H3N2 Day 29 | 90 | 91
  B/Victoria Day 1 | 32 | 41
  B/Victoria Day 29 | 76 | 80
  B/Yamagata Day 1 | 37 | 40
  B/Yamagata Day 29 | 84 | 81

21. Secondary Outcome: Number of Participants With Local and Systemic Adverse Events (AEs)
Description: Systemic AEs: fatigue, headache, myalgia, arthralgia, nausea, dizziness, chills, and fever. Solicited local (injection site) AEs: injection site pain, erythema, and swelling. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 8 and Day 36 (up to 7 days after each study vaccination)
Population: Safety Analysis Set (SAF), which included all participants in the Exposed Set (participants who received at least one dose of a study vaccine) who provided any evaluable post-vaccination reactogenicity and/or safety data. Number analyzed = participants evaluable at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV | Cohort A Group 3a: QIV + Placebo + ARCT-2303 | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV | Cohort B Group 3b: aQIV + Placebo + ARCT-2303
Number analyzed (Participants) | 403 | 403 | 398 | 99 | 98 | 98
Participants
  Solicited Local AE after First Vaccination (up to Day 8) | 283 | 296 | 167 | 41 | 30 | 20
  Solicited Systemic AE after First Vaccination (up to Day 8) | 255 | 258 | 162 | 36 | 23 | 25
  Solicited Local AE after Second Vaccination (up to Day 36): number analyzed (Participants) | 393 | 394 | 390 | 95 | 97 | 96
  Solicited Local AE after Second Vaccination (up to Day 36) | 38 | 146 | 263 | 5 | 15 | 22
  Solicited Systemic AE after Second Vaccination (up to Day 36): number analyzed (Participants) | 393 | 394 | 390 | 95 | 97 | 96
  Solicited Systemic AE after Second Vaccination (up to Day 36) | 105 | 118 | 217 | 14 | 15 | 17

22. Secondary Outcome: Number of Participants With Unsolicited AEs
Description: An unsolicited AE was an AE that was not listed as 'solicited' and was defined as any spontaneously occurring AE (serious and non-serious). Potential unsolicited AEs may have been medically attended (defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a healthcare provider) or were of concern to the participants. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to Day 29 (Up to 28 days after first study vaccination) and up to Day 57 (28 days after second study vaccination)
Population: Safety Analysis Set, which included all participants in the Exposed Set (participants who received at least one dose of a study vaccine) who provided any evaluable post-vaccination reactogenicity and/or safety data. Overall number of participants analyzed = participants evaluable for the outcome measure. Number analyzed = participants evaluable at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV | Cohort A Group 3a: QIV + Placebo + ARCT-2303 | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV | Cohort B Group 3b: aQIV + Placebo + ARCT-2303
Number analyzed (Participants) | 403 | 403 | 398 | 99 | 98 | 98
Participants
  Day 29 | 79 | 81 | 68 | 13 | 8 | 16
  Day 57: number analyzed (Participants) | 393 | 394 | 390 | 95 | 97 | 96
  Day 57 | 71 | 62 | 75 | 9 | 6 | 17

23. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), AEs Leading to Early Termination From Study, Medically Attended Adverse Event (MAAEs), and Adverse Event of Special Interest (AESIs)
Description: SAEs were defined as any event that resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly or birth defect, or was an important medical event. A MAAE was an AE that led to an unscheduled visit (including a telemedicine visit) to a healthcare practitioner. AESIs were defined as AEs potentially associated with Coronavirus Disease 2019 (COVID-19) and COVID-19 vaccines. Number of participants with AEs leading to early termination included AEs leading to death. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 up to Day 181
Population: Safety Analysis Set, which included all participants in the Exposed Set (participants who received at least one dose of a study vaccine) who provided any evaluable post-vaccination reactogenicity and/or safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV | Cohort A Group 3a: QIV + Placebo + ARCT-2303 | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV | Cohort B Group 3b: aQIV + Placebo + ARCT-2303
Number analyzed (Participants) | 403 | 403 | 398 | 99 | 98 | 98
Participants
  SAEs | 7 | 5 | 6 | 2 | 3 | 5
  AEs Leading to Early Termination from Study | 0 | 1 | 0 | 0 | 0 | 1
  MAAEs | 103 | 95 | 100 | 19 | 13 | 19
  AESIs | 1 | 1 | 3 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 181
Description: Safety analysis set, which included all participants in the Exposed Set (all participants who received at least one dose of a study vaccine in this study) who provided any evaluable post-vaccination reactogenicity and/or safety data. As pre-specified, mortality and adverse event data were collected and reported for participants enrolled in this study. The historical control group were not considered enrolled and were not assessed for deaths/adverse events in this study.
Arm/Group | Cohort A Group 1a: ARCT-2303+ QIV + Placebo | Cohort A Group 2a: ARCT-2303 + Placebo + QIV | Cohort A Group 3a: QIV + Placebo + ARCT-2303 | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV | Cohort B Group 3b: aQIV + Placebo + ARCT-2303
All-Cause Mortality (participants affected / at risk) | 0/403 | 0/403 | 0/398 | 0/99 | 0/98 | 1/98
Serious Adverse Events (participants affected / at risk) | 7/403 | 5/403 | 6/398 | 2/99 | 3/98 | 5/98
Other Adverse Events (participants affected / at risk) | 65/403 | 59/403 | 49/398 | 6/99 | 0/98 | 14/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort A Group 1a: ARCT-2303+ QIV + Placebo (N=403) | Cohort A Group 2a: ARCT-2303 + Placebo + QIV (N=403) | Cohort A Group 3a: QIV + Placebo + ARCT-2303 (N=398) | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo (N=99) | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV (N=98) | Cohort B Group 3b: aQIV + Placebo + ARCT-2303 (N=98)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myopericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malignant glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 3 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/259 | 1/255 | 0/243 | 0/64 | 0/68 | 0/63 — "At risk" values have been updated since this is a sex-specific event.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A Group 1a: ARCT-2303+ QIV + Placebo (N=403) | Cohort A Group 2a: ARCT-2303 + Placebo + QIV (N=403) | Cohort A Group 3a: QIV + Placebo + ARCT-2303 (N=398) | Cohort B Group 1b: ARCT-2303 + Adjuvanted QIV (aQIV) + Placebo (N=99) | Cohort B Group 2b: ARCT-2303 + Placebo + aQIV (N=98) | Cohort B Group 3b: aQIV + Placebo + ARCT-2303 (N=98)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
COVID-19 (Infections and infestations) | 22 | 21 | 18 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 43 | 38 | 31 | 3 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 5
Hypertensive urgency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT06279871/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT06279871/SAP_001.pdf